CLINICAL TRIAL: NCT03021135
Title: Conventional Endoscopic Mucosal Resection (With Submucosal Injection) Versus Underwater Endoscopic Mucosal Resection (Without Submucosal Injection) for Colorectal Non-pedunculated Colorectal Lesions
Brief Title: Conventional Endoscopic Mucosal Resection vs Underwater Resection for Colorectal Non-pedunculated Colorectal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 941/16
Record Dates: First submitted 2016-11-04; First posted 2017-01-13 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2022-04

CONDITIONS: Adenoma; Colorectal Neoplasms
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Mucosal Resection (Active Comparator): C-EMR will be made with saline injection with the indigo carmine.
  Interventions: Procedure: Conventional Endoscopic Mucosal Resection
- Underwater Mucosal Resection (Experimental): UW-EMR will be made after the complete filling of lumen with water.
  Interventions: Procedure: Underwater Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Conventional Endoscopic Mucosal Resection — Conventional Endoscopic Mucosal Resection
  Other Names: EMR
  Arms: Conventional Mucosal Resection
Procedure: Underwater Endoscopic Mucosal Resection — Underwater Endoscopic Mucosal Resection
  Other Names: U-EMR
  Arms: Underwater Mucosal Resection

SUMMARY:
Randomized, comparative and prospective study between Conventional Endoscopic Mucosal Resection for the removal of flat or sessile colorectal lesions without previous attempt to resection.

DETAILED DESCRIPTION:
This prospective randomized trial was conducted in 2 academic services: Instituto do Câncer do Estado de São Paulo and Centro de Diagnóstico em Gastroenterologia, both linked to the University of São Paulo. The clinical study was performed in accordance to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years with sessile or flat Colorectal Lesions (measuring between 10 and 40mm), who consent to this study

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients with pedunculated, depressed or mixed lesions.
* Patients with lesions smaller than 10 mm or larger than 40 mm.
* Patients with lesions that are inflammatory, neuroendocrine or stromal at the pathology.
* Patients with lesions that were submitted to prior attempt to endoscopic resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Technical success rate | three years
Safety (incidence of complications); | three years
Local recurrence. | Four years

SECONDARY OUTCOMES:
Resection rate en bloc | three years
Time of resection | Three years
Sydney resection ratio (characterized by the following equation - lesion size in millimeters | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Lenz, PhD, Principal Investigator — Cancer Institute of the state of São Paulo (ICESP)
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results — http://doi.org/10.1016/j.gie.2022.10.033